CLINICAL TRIAL: NCT05069740
Title: Mechanisms and Interventions Addressing Accelerated Cardiovascular Disease Risk in Endometriosis
Brief Title: Endometriosis and Microvascular Dysfunction: Role of Inflammation
Acronym: Endo3/SA2
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Lacy Alexander, Professor of Kinesiology, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 18369
Record Dates: First submitted 2021-09-10; First posted 2021-10-06 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Endometriosis
Keywords: skin blood flow; inflammation; Lectin-like oxidized LDL receptor (LOX-1); intradermal microdialysis
MeSH Terms: conditions — Endometriosis; Inflammation | interventions — salicylsalicylic acid

STUDY DESIGN:
Intervention Model Description: This is a single blind placebo controled cross over study. Two groups of women complete this study: 1) healthy women between the ages of 18 and 45 years (Controls); 2) women between the ages of 18 and 45 years with endometriosis. Once consented and screening, each subject is randomized to either 5 days of salsalate or placebo. On day 5, each subject participates in a cutaneous microdialysis (MD) and flow mediated dilation (FMD) experiment. After a 2-week washout, the participant returns to repeat the study with the other oral drug (salsalate/placebo). These treatments are blinded to only the investigators. The participants and nurse on staff knows which treatment the subject is taking if there are any questions or safety concerns.
Who Masked: Investigator
Masking Description: These treatments/placebo are blinded to the investigators. The subjects, physician, and the nurse on staff knows which treatment the subject is taking if there are any questions or safety concerns.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Salsalate (Experimental): 3000 mg/day salsalate (1500 mg twice daily) for 5 days
  Interventions: Drug: Salsalate Pill
- Placebo (Placebo Comparator): 1 capsule contain microcrystalline cellulose filler (twice daily) for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salsalate Pill — Salsalate acts as an NFkB inhibitor to reduce systemic inflammation
  Arms: Salsalate
Drug: Placebo — Placebo for the salsalate intervention
  Arms: Placebo

SUMMARY:
The purpose of this study is to better understand the underlying mechanisms associated with elevated cardiovascular disease risk in women with endometriosis, and to measure the effectiveness of emerging endometriosis treatments on outcomes specific to cardiovascular dysfunction.

Epidemiologic data demonstrate a clear association between endometriosis, reproductive risk factors, inflammation and cardiovascular (CV) risk. Circulating factors, low-density lipoprotein (LDL) and oxidized LDL (oxLDL), are two of many biomarkers of cardiovascular and inflammatory disease of endometriosis. An important signaling mechanism through which circulating LDL and oxLDL act is the lectin-like oxidized LDL receptor (LOX-1). LOX-1 signal transduction functionally results in pronounced endothelial dysfunction, a hallmark of CV. The investigators hypothesis that one factor mediating the elevated risk of cardiovascular disease in endometriosis is systemic inflammation and activation of LOX-1 receptor mechanisms.

DETAILED DESCRIPTION:
Endometriosis is an estrogen-dependent gynecological disorder associated with considerable chronic pelvic pain, pain during intercourse, and is a major cause of infertility. This disorder affects 6% - 10% of reproductive age women and can be as high as 35-50% in women experiencing pain or infertility. Endometriosis derives from the presence of endometrium-like tissue in sites outside the uterine cavity. While endometriosis is a local inflammatory syndrome, the inflammatory process is systemic.

Endometriosis is associated with higher risk of hypercholesterolemia and hypertension 8. Epidemiologic data demonstrate a clear association between endometriosis, reproductive risk factors, inflammation and cardiovascular (CV) risk.

Endometriosis a disease of inflammation and increased systemic inflammatory cytokine production, although the precise mechanisms by which localized lesion results in systemic inflammation are incompletely understood. Published data confirm an elevation of several inflammatory cytokines in the circulation of women with endometriosis. Alterations in circulating miRNAs specific to endometriosis are one mechanism causing immune dysfunction and subsequent increased cytokine expression in areas remote from the endometriotic lesions. This aberrant increase in systemic cytokine production is a highly plausible putative link to accelerated vascular dysfunction and atherosclerosis in women with endometriosis.

The circulating factors LDL and oxidized LDL are two of the many biomarkers of cardiovascular and inflammatory disease of endometriosis. An important signaling mechanism through which circulating LDL and oxLDL act is the lectin-like oxidized LDL receptor (LOX-1). LOX-1 is a ubiquitously expressed scavenger receptor, stimulated by oxLDL, Ang II, and other inflammatory cytokines, and inhibited by estrogen. LOX-1 is the upstream signaling initiator of mechanisms including increased oxidant production, reduced nitric oxide (NO) metabolism, and impaired intracellular trafficking. Thus, LOX-1 signal transduction functionally results in pronounced endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women between the ages of 18 and 45 years (Controls), taking oral contraceptive or with regular menses every 26-34 days
* Women between the ages of 18 and 45 years with endometriosis (diagnosis by prior laparoscopy by subject's own physician <5 years prior, and reported by the subject to the researchers)
* Tylenol if the subject has acute pain is allowed
* Contraceptive use is allowed

Exclusion Criteria:

* Use of nicotine-containing products (e.g. smoking, chewing tobacco, etc.)
* Diabetes (HbA1C 6.5%)
* BP>140/90
* Taking pharmacotherapy that could alter peripheral vascular control (e.g. insulin sensitizing, cardiovascular medications)
* Pregnancy
* Breastfeeding
* Taking illicit and/or recreational drugs
* Abnormal liver function
* Rash, skin disease, disorders of pigmentation, known skin allergies
* Diagnosed or suspected metabolic or cardiovascular disease
* Persistent unexplained elevations of serum transaminases
* Known allergy to latex or investigative substances (including salsalate or simvastatin)
* History of gastrointestinal bleeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
cutaneous vascular conductance | 5 days after treatment
  doppler flowmetry used to measure cutaneous vascular conductance (cvc = red cell flux/mean arterial pressure) to assess microvascular endothelial function
brachial artery diameter and blood flow velocity | 5 days after treatment
  continuous ultrasound imaging measurements of brachial artery diameter and blood flow velocity to assess endothelial function
Sera LOX-1 protein expression | 5 days after treatment
  Peripheral Blood Mononuclear Cell Isolation, LOX-1 expression quantified using real time pCR
Biopsy LOX-1 protein expression | 5 days after treatment
  Bio-Rad DC assay, western blot technique used for LOX-1 protein receptor expression

SECONDARY OUTCOMES:
sera reproductive hormone analysis | 5 days after treatment
  analysis of plasma estradiol, progesterone, and sex hormone binding globulin determined through hormone assay
sera cytokine expression analysis | 5 days after treatment
  expression of cytokines CRP, TNF-a, IL-1B, IL-6, IL-8 determined through multiplex assay
skin biopsy biochemical analysis | 5 days after treatment
  the expression of estrogen receptor alpha and beta, the protein pVASP/VASP, and the enzyme peNOS/eNOS is determined using Bio-Rad DC assay, western blot technique

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No